CLINICAL TRIAL: NCT02031107
Title: Randomized Controlled Trial of Transcranial Theta-burst Stimulation and Transcranial Direct Current Stimulation in Subacute Stroke
Brief Title: Randomized Trial of Transcranial Theta-burst Stimulation and Transcranial Direct Current Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adrian Guggisberg (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor-Investigator, Adrian Guggisberg, Médecin adjoint agrégé, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SNF-146639-1
Record Dates: First submitted 2014-01-06; First posted 2014-01-09 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Stroke
Keywords: stroke; brain stimulation; electroencephalography; functional magnetic resonance imaging; functional connectivity
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- cTBS (Active Comparator): A transcranial magnetic stimulator (MagPro X100, Medtronic Functional Diagnostics, Skovlunde, Denmark) will deliver continuous bursts of bipolar magnetic pulses exerting an inhibition on the underlying brain tissue (cTBS). The stimulation coil will be placed over the unaffected primary motor cortex. The stimulation protocol implies 200 bursts, each consisting of three pulses applied at 30 Hz, repeated at inter-burst intervals of 167 ms. Two stimulation trains of 30 s, separated by 15 min, will be applied 3 times per week for 3 weeks and will be immediately followed by physical therapy.
  Interventions: Device: cTBS
- cathodal tDCS (Active Comparator): A stimulator (NeuroConn GmbH, Illmenau, Germany) will deliver cathodal transcranial direct current stimulation (tDCS) of the unaffected motor cortex. The anode will be placed over the contralateral supraorbital region. Stimulation will be performed for 25 min, 3 times per week for 3 weeks during upper extremity treatment sessions.
  Interventions: Device: cathodal tDCS
- sham stimulation (Sham Comparator): This group will receive the same stimulation protocol as used for the active groups except that sham stimuli will be applied. Half of the patients receive sham cTBS, the other half sham tDCS.
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: cTBS
  Other Names: MagPro X100
  Arms: cTBS
Device: cathodal tDCS
  Other Names: NeuroConn
  Arms: cathodal tDCS
Device: sham stimulation
  Arms: sham stimulation

SUMMARY:
Background: Stroke is a leading cause of adult disability. Non-invasive brain stimulation can induce significant and sustained improvements in functional outcome. However the effect is inconsistent and difficult to predict, in particular in the subacute phase after stroke. Although several different stimulation techniques are available, it is unknown which is suitable for which patient.

Objectives: This study has three main objectives:

1. To compare the effects of two techniques of non-invasive brain stimulation (cTBC, continuous theta-burst stimulation; tDCS, direct current transcranial stimulation) on clinical recovery in patients with subacute stroke.
2. To assess the effect of these brain stimulation techniques on brain organization with non-invasive imaging.
3. To find clinical and neural predictors of responsiveness to brain stimulation therapy.

Method: 45 patients with ischemic or hemorrhagic stroke will be randomly assigned to one of 3 groups: cTBS, tDCS, or sham stimulation. Each group will receive the corresponding stimulation therapy 3 times per week for 3 weeks, immediately before intensive physical therapy. Before and after the treatment period, standardized assessments of sensorimotor function areas are obtained together with electroencephalography and functional magnetic resonance recordings. These recordings will be used to analyze and compare the neural effects of each treatment modality.

Clinical Implication: The results of this study might help optimize and individualize stimulation treatment for patients with subacute stroke. It may hence facilitate the transfer of brain stimulation therapy to routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* ischemic or hemorrhagic stroke leading to unilateral deficits in motor function with significant impact on independence and daily activities at the beginning of rehabilitation
* less than 10 weeks after stroke onset.

Exclusion Criteria:

* epileptic seizures
* metallic objects in the brain
* presence of implants or neural stimulators
* pregnancy
* sleep deprivation
* recent traumatic brain injury
* delirium or disturbed vigilance
* inability to participate in 1h treatment sessions
* severe language comprehension deficits
* skull breach
* new stroke lesions during rehabilitation
* medical complications

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in compound motor score slope at week 4 | week 4 after treatment start
  The Fugl Meyer motor assessment (FMA), the Nine Hole Peg test (expressed as pegs per minute), and the Jamar dynamometer strength of the affected arm are normalized to the healthy arm and averaged to a compound motor score. This score is obtained twice before treatment (at weeks -1 and 0 relative to treatment start), and twice after treatment (at weeks 4 and 8). Primary outcome measure is the change in slope from week 0 to 4 as compared to the slope between week -1 and 0.
Change in alpha-band coherence between the affected motor cortex and the rest of the brain | Week 4
  Calculated from electroencephalography recordings

SECONDARY OUTCOMES:
Change in Fugl Meyer Upper Extremity Motor Score at week 4 | Week 4
Change in Fugl Meyer Upper Extremity Motor Score at week 8 | Week 8
Change in alpha-band coherence between the unaffected motor cortex and the rest of the brain | Week 4
Change in activity of daily life scale (motor activity log, MAL) | Week 4
Change in activity of daily life scale (motor activity log, MAL) | Week 8
Number of adverse events | Week 4
Number of adverse events | Week 8

OTHER OUTCOMES:
Total Fugl Meyer motor assessment score at week 4 | Week 4
Total Fugl Meyer motor assessment score at week 8 | Week 8
Change in average velocity in the Nine Hole Peg test at week 4 | Week 4
  expressed in pegs/sec
Change in average velocity in the Nine Hole Peg test at week 8 | Week 8
  expressed in pegs/sec
Change in Jamar Dynamometer strength at week 4 | Week 4
Change in Jamar Dynamometer strength at week 8 | Week 8
Change in Score of the Box and Block test, week 4 | Week 4
Change in Score of the Box and Block test, week 8 | week 8
Correlation between change in alpha band coherence and clinical improvements | Week 4
  Alpha band coherence is calculated from electroencephalography (EEG) recordings
Change in fractional anisotropy of the affected cortico-spinal tract | Week 4
  Calculated from diffusion tensor imaging (DTI) sequences of magnetic
Change in correlations of spontaneous fMRI fluctuations within the motor network | Week 4
  Calculated from functional magnetic resonance (fMRI) recordings

CONTACTS AND LOCATIONS:
Overall Officials: Adrian G Guggisberg, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Service de Neurorééducation, Unversity Hospital, Geneva, Switzerland

REFERENCES:
- [Background] Rizk S, Ptak R, Nyffeler T, Schnider A, Guggisberg AG. Network mechanisms of responsiveness to continuous theta-burst stimulation. Eur J Neurosci. 2013 Oct;38(8):3230-8. doi: 10.1111/ejn.12334. Epub 2013 Aug 14. PMID 23941616
- [Derived] Nicolo P, Magnin C, Pedrazzini E, Plomp G, Mottaz A, Schnider A, Guggisberg AG. Comparison of Neuroplastic Responses to Cathodal Transcranial Direct Current Stimulation and Continuous Theta Burst Stimulation in Subacute Stroke. Arch Phys Med Rehabil. 2018 May;99(5):862-872.e1. doi: 10.1016/j.apmr.2017.10.026. Epub 2017 Dec 7. PMID 29223708